CLINICAL TRIAL: NCT06474533
Title: Fluoroethyltyrosine for the Evaluation of Intracranial Neoplasm
Status: Recruiting | Type: Observational
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Co-Principal Investigator, IND Holder, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: 24924; NCI-2024-04996 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Intracranial Neoplasm
Keywords: Imaging Studies
MeSH Terms: conditions — Brain Neoplasms | interventions — Fluorine-18; (18F)fluoroethyltyrosine; O-(2-fluoroethyl)tyrosine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population 1: Participants with intracranial neoplasms: Participants with intracranial neoplasms (glial or metastatic disease) with concern for recurrence or progression on conventional imaging.
  Interventions: Drug: Fluorethyltyrosine (18-F); Procedure: Positron Emission Tomography (PET)
- Population 2: Participants with suspected glial neoplasms: Participants with suspected glial neoplasms (Grade 2 - 4) planning to undergo biopsy or surgery prior to non-investigational, standard-of-care, primary treatment (radiation therapy and/or surgery)
  Interventions: Drug: Fluorethyltyrosine (18-F); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: Fluorethyltyrosine (18-F) — Given intravenously (IV)
  Other Names: Fluoroethyltyrosine (FET); FET; O-(2-[18F]fluoroethyl)-L-tyrosine (FET)
Procedure: Positron Emission Tomography (PET) — Undergo Imaging Procedure
  Other Names: PET scan; PET

SUMMARY:
This is a single center study investigating the use of Fluoroethyltyrosine (FET) in the detection of brain tumors. FET accumulates in malignant cells within intracranial neoplasms and can be used to detect recurrent disease and characterize grade of glial neoplasms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To determine if FET Positron Emission Tomography (PET) scan can differentiate between benign treatment-related changes and recurrence in comparison to pathology in population 1 with recurrent metastatic disease and high-grade gliomas.
2. To determine if FET PET scan can differentiate between low-grade and high-grade gliomas in population 2.

SECONDARY OBJECTIVES:

1. To determine if FET PET scan can differentiate between benign treatment- related changes and recurrence in comparison to pathology or imaging follow-up in population 1.
2. To determine if FET PET scan can differentiate between benign treatment- related changes and recurrence in comparison to pathology in population 1 with recurrent low-grade gliomas.

EXPLORATORY OBJECTIVES:

1. To assess relationships between serial FET PET scan and clinical outcome in population 1 with recurrent metastatic disease and gliomas.

OUTLINE:

Participants will receive a single PET scan lasting for about 40 minutes in an outpatient setting after an injection with FET. Adult participants may undergo up to two repeat FET PET scans. Adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Presence or suspicion of intracranial neoplasm in two populations:

  * Population 1: Participants after primary treatment (radiation therapy and/or surgery) with suspicion of recurrence on MRI.
  * Three sub-populations will be considered:

    * Recurrent metastatic lesions.
    * Recurrent high-grade gliomas (Grades 3 and 4).
    * Recurrent low-grade gliomas (Grade 2).
  * Population 2: Participants prior to primary treatment with planned biopsy or surgical resection.
* Age > 3 years.

Participants in other clinical trials will be eligible for this study including patients undergoing surgery guided by 5-aminolevulinic acid.

Exclusion Criteria:

* Participants with known incompatibility to PET or Computerized tomography (CT)/magnetic resonance imaging (MRI) scans.
* Participants unlikely to comply with study procedures, restrictions and requirements and judged by the Investigator to be unsuitable for study participation.

  * Sedation or anesthesia can be used for participants who cannot tolerate the exam.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children over the age of 3 with intracranial neoplasms (glial or metastatic disease).
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Intracranial lesion tumor-to-background ratio (TBRmax) | Up to 3 years
  The maximum TBR (TBRmax) will be calculated by dividing the SUVmean of the 1.6 centimeter (cm) diameter circular region of interest (ROI) by the mean standardized uptake value (SUVmean) of background normal tissue.
Percentage of accurate prediction of presence of tumor (Population 1) | Up to 3 years
  The percentage of radiological read responses that accurately predict the presence of recurrent tumor in patients previously treated with surgery and/or radiation for population 1, broken down by metastatic disease, high-grade gliomas and low-grade gliomas will be reported
Percentage of radiological read responses | Up to 3 years
  The percentage of radiological reads with a binary characterization of scan study as positive for recurrence disease in population 1, and positive for high-grade glial neoplasm in population 2 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Villanueva-Meyer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No